CLINICAL TRIAL: NCT02554123
Title: Reduction of Postoperative Pain and Improvement of Patients´Comfort After Milligan-Morgan Haemorrhoidectomy With Application of Vitamin E Ointment
Brief Title: Reduction of Postoperative Pain After Milligan-Morgan Haemorrhoidectomy With Application of Vitamin E Ointment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRJC15-22
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin E ointment (Experimental): Vitamin E ointment application. Every 12 hours during 7 days.
  Interventions: Drug: Vitamin E ointment application
- Vaseline ointment (Placebo Comparator): Vaseline ointment application. Every 12 hours during 7 days.
  Interventions: Drug: Vaseline ointment application

INTERVENTIONS:
Drug: Vitamin E ointment application — Vitamin E ointment application. Every 12 hours during 7 days.
  Arms: Vitamin E ointment
Drug: Vaseline ointment application — Vaseline ointment application. Every 12 hours during 7 days.
  Arms: Vaseline ointment

SUMMARY:
A prospective ranfomized clinical study of patients undergoing Milligan Morgan´s haemorrhoidectomy at Hospital Universitario Rey Juan Carlos (Móstoles-Spain) will be performed. The patients will be randomized into 2 groups:

* Experimental group (EG): Patients undergoing Milligan Morgan´s procedure and application of Vitamin E ointment on the surgical bed.
* Control group (CG): Patients undergoing Milligan Morgan´s procedure and application of Vaseline on the surgical bed.

Postoperative pain determined by VAS at the 1st, 3rd and 7th postoperative days, and need for morphine rescue will be investigated.

DETAILED DESCRIPTION:
A prospective ranfomized clinical study of patients undergoing Milligan Morgan´s haemorrhoidectomy at Hospital Universitario Rey Juan Carlos (Móstoles-Spain) will be performed. The patients will be randomized into 2 groups:

* Experimental group (EG): Patients undergoing Milligan Morgan´s procedure and application of Vitamin E ointment on the surgical bed.
* Control group (CG): Patients undergoing Milligan Morgan´s procedure and application of Vaseline on the surgical bed.

Postoperative pain determined by VAS at the 1st, 3rd and 7th postoperative days, and need for morphine rescue will be investigated by a blined epidemiology nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Milligan Morgan´s haemorrhoidectomy at Hospital Universitario Rey Juan Carlos (Móstoles-Spain).
* Haemorrhoids grade III and IV
* The patients sign an Informed Consent Form agreeing their participation in the study.

Exclusion Criteria:

* Patients undergoing other surgical techniques for haemorrhoidectomy, different tan Milligan Morgan
* Haemorrhoids grade I and II
* Patients with medical or surgical pathologies that do not allow the participation in the study
* Disability to understand and accept the entry in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | From the first to the 7th postoperative days
  Postoperative pain will be quantified with a VAS scale at the 1st, 3rd and 7th postoperative days

SECONDARY OUTCOMES:
Need for morphine rescue | 24 hours after surgery
  Need for morphine rescue will be quantified in the first 24 hours after surgery during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Duran, MD, PhD, Study Director — Hospital Rey Juan Carlos